CLINICAL TRIAL: NCT00001112
Title: A Phase I Study To Determine the Safety of the Optimal Monocyte Activating Administration Schedule of Subcutaneous Human Recombinant Interferon-gamma in ZDV-Treated Patients With AIDS
Brief Title: The Safety and Effectiveness of Injections of Human Recombinant Interferon-gamma in Patients With AIDS Who Have Taken Zidovudine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 072; 11046 (Registry Identifier: DAIDS ES Registry ID)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Monocytes; Interferon-gamma, Recombinant; Injections, Subcutaneous; Immune System; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Blood Bactericidal Activity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; interferon gamma-1b

INTERVENTIONS:
Drug: Zidovudine
Drug: Interferon gamma-1b

SUMMARY:
To find out which of four doses of (recombinant) human interferon gamma (IFN-G) is most effective in stimulating the white blood cells (monocytes) to fight infection and to see if treatment with IFN-G can strengthen the ability of AIDS patients to control infections. This study will also determine how long after a single injection of IFN-G white blood cells remain stimulated.

AIDS is a disease that progressively destroys that aspect of the body's defense called the immune system. It is particularly harmful to a class of cells called helper T-lymphocytes. The specific opportunistic infections and malignancies associated with AIDS have been treated with therapies that are often poorly tolerated by the patients and are associated with dose-limiting toxicities. The principal focus of AIDS therapy research at present is to control the underlying retroviral infection and to restore immune function with recombinant lymphokines, adoptive immunotherapy, and/or lymphocyte transplants. These treatments include zidovudine (AZT), which has been shown to control the HIV infection, and IFN-G, a lymphokine which activates tumor-destroying and germ-killing functions. Studies are needed to find the dose by which IFN-G works best.

DETAILED DESCRIPTION:
AIDS is a disease that progressively destroys that aspect of the body's defense called the immune system. It is particularly harmful to a class of cells called helper T-lymphocytes. The specific opportunistic infections and malignancies associated with AIDS have been treated with therapies that are often poorly tolerated by the patients and are associated with dose-limiting toxicities. The principal focus of AIDS therapy research at present is to control the underlying retroviral infection and to restore immune function with recombinant lymphokines, adoptive immunotherapy, and/or lymphocyte transplants. These treatments include zidovudine (AZT), which has been shown to control the HIV infection, and IFN-G, a lymphokine which activates tumor-destroying and germ-killing functions. Studies are needed to find the dose by which IFN-G works best.

Patients, who may participate in all three parts of the study, are maintained on a stable dose of AZT. In part A (optimal dose), five AIDS patients who have had an AIDS related opportunistic infection receive 4 once-weekly increasing doses of IFN-G. Monocyte antimicrobial activity is examined in test tube studies before and after each injection of IFN-G. In part B, five patients receive the optimal dose of IFN-G established in part A. Patients enrolled from part A have completed at least 2 weeks of part A before enrolling in part B. Antimicrobial activity is examined 1, 2, and 3 days after a single injection of the optimal dose of IFN-G (determined in part A). In part C (safety and tolerance of combined treatment of IFN-G and AZT), patients are treated with IFN-G for 4 weeks using the optimal dose and administration schedule derived from parts A and B.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylactic antibiotics.
* Tylenol (650 mg orally every 6 hours as needed for temperature > 38.5 degrees C).
* Meperidine (25 - 50 mg intravenously, once, for severe rigors if systolic blood pressure is > 90 mmHg).

Patients must meet criteria for AIDS classification (CDC) category IV C-1.

* Patients must have had one or more prior opportunistic infections identified in surveillance definition of AIDS. Patients whose AIDS-defining illness is Kaposi's sarcoma are also eligible if they have previously had one of the secondary infectious diseases identified in category C-1.

Prior Medication:

Required:

* Patients must have been receiving zidovudine (AZT) on a stable dosage regimen for at least 8 weeks immediately preceding entry into study.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Clinically significant cardiac (= or > class II, New York Heart Association) or peripheral vascular disease that requires treatment.
* Presence of an active opportunistic infection that requires treatment.
* Hemorrhagic diathesis or active bleeding disorder.
* Clinically apparent vascular disease.

Concurrent Medication:

Excluded:

* Medications required for treatment of active cardiac disease.
* Ongoing therapy with anticoagulants or thrombolytic agents.

Patients with the following are excluded:

* Clinically significant cardiac (= or > class II, New York Heart Association) or peripheral vascular disease that requires treatment.
* Presence of an active opportunistic infection that requires treatment.
* Hemorrhagic diathesis or active bleeding disorder.
* Clinically apparent vascular disease.

Prior Medication:

Excluded within 4 weeks of study entry:

* Antiviral chemotherapy other than zidovudine.
* Excluded within 12 weeks of study entry:
* Immunosuppressive or cytotoxic therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Study Completion 1993-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: HW Murray, Study Chair
Locations (1):
- Cornell University A2201, New York, New York, United States

REFERENCES:
- [Background] Murray HW, Scavuzzo D, Jacobs JL, Kaplan MH, Libby DM, Schindler J, Roberts RB. In vitro and in vivo activation of human mononuclear phagocytes by interferon-gamma. Studies with normal and AIDS monocytes. J Immunol. 1987 Apr 15;138(8):2457-62. PMID 3104467